CLINICAL TRIAL: NCT01412970
Title: Non-invasive Measurement of Central Hemodynamics and Heart-lung Interactions by Electrical Impedance Tomography
Brief Title: Non-invasive Measurement of Central Hemodynamics by Electrical Impedance Tomography
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: received no funding
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry); Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DFG3171_2-1
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Comparison of Availability for Prediction of Volume Responsiveness; Comparison of Limits of Agreement for Invasive and Non-invasive Measurement of Stroke Volume Variation
Keywords: hemodynamic monitoring; volume responsiveness; electrical impedance tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study group (Other): comparison of ability to predict volume responsiveness and precision of measurement of stroke volume variation assessed by electrical impedance tomography in comparison to clinically established invasive hemodynamic monitoring devices, i.e. arterial pulse contour analysis during volume loading procedures
  Interventions: Other: volume loading

INTERVENTIONS:
Other: volume loading — volume loading according to functional parameters of cardiac preload, i.e. stroke volume variations measured by arterial pulse contour analysis

SUMMARY:
The purpose of this study is to evaluate the ability to measure central hemodynamics and heart-lung interactions non-invasively by electrical impedance tomography and compare it to clinically established hemodynamic monitoring.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the ability to measure central hemodynamics and heart-lung interactions non-invasively by electrical impedance tomography and compare it to clinically established hemodynamic monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Indication for advanced invasive hemodynamic monitoring due to operative procedure
* Necessity of postoperative invasive ventilation

Exclusion Criteria:

* Age <18 years
* known affections cardiac function
* presence of cardiac arrhythmias
* contraindication for placement of central venous or femoral artery catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Estimated); Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Ability to assess volume responsiveness by electrical impedance tomography | within 3 hrs after surgical procedure
  Assessment of volume responsiveness by electrical impedance tomography in mechanically ventilated patients by measurement of stroke volume variations under stepwise volume loading

SECONDARY OUTCOMES:
precision of estimation of non invasive measurement of stroke volume variation | within 3 hours after surgery
  precision of estimation of non invasive measurement of stroke volume variation by electrical impedance tomography in comparison to clinically established, invasive advanced hemodynamic monitoring devices

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Reuter, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Maisch S, Bohm SH, Sola J, Goepfert MS, Kubitz JC, Richter HP, Ridder J, Goetz AE, Reuter DA. Heart-lung interactions measured by electrical impedance tomography. Crit Care Med. 2011 Sep;39(9):2173-6. doi: 10.1097/CCM.0b013e3182227e65. PMID 21666450